CLINICAL TRIAL: NCT03443453
Title: A Single-Center, Randomised, 4-Period, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability, and Effect of Food on Pharmacokinetics Following Single Doses of MIV-711 Capsule and Tablet Formulations in Healthy Volunteers
Brief Title: A Bioavailability Study of MIV-711 Oral Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MIV-711-102
Record Dates: First submitted 2018-01-22; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — MIV-711

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MIV-711 ABCD (Experimental): Subjects will first receive the tablet formulation under fasted conditions (A) followed by the tablet formulation administered under fed conditions (B). Thereafter they will receive the capsule formulation under fasted conditions (C) followed by the capsule formulation administered under fed conditions (D).
  Interventions: Drug: MIV-711
- MIV-711 CDAB (Experimental): Subjects will first receive the capsule formulation under fasted conditions (C)followed by the capsule formulation administered under fed conditions (D). Thereafter they will receive the tablet formulation under fasted conditions (A) followed by the tablet formulation administered under fed conditions (B).
  Interventions: Drug: MIV-711

INTERVENTIONS:
Drug: MIV-711 — MIV-711 administered as tablets and capsules at four occasions

SUMMARY:
This is a single-Center, Randomised, 4-Period, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability, and Effect of Food on Pharmacokinetics following Single Doses of MIV-711 Capsule and Tablet Formulations in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria (subset):

* Healthy, adult, male or female, 19-55 years of age, inclusive, at screening.
* Body mass index (BMI) ≥ 18.5 and ≤ 30.0 kg/m2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
* If not a menopausal female or surgically sterile male or female, subjects must be willing to practice at least one of the in the CSP described highly effective methods of birth control for at least a (partner's) menstrual cycle before and for 3 months after study drug administration.
* For a female of non-childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

  * hysteroscopic sterilization;
  * bilateral tubal ligation or bilateral salpingectomy;
  * hysterectomy;
  * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 2 years prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.

Exclusion Criteria (subset):

* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, that could affect the action, absorption, or disposition of MIV-711 or may confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of known structural cardiac abnormalities, syncope, cardiac conduction problems (first, second, or third degree heart blocks, bundle branch block, or incomplete block, atrial fibrillation and/or paroxysmal atrial fibrillation, sick sinus syndrome or prolonged QTc interval), inappropriate sinus bradycardia, deviant ECG morphology or exercise related cardiac events.
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study. Medication listed as part of acceptable birth control methods will be allowed.
  * Any drugs known to be inducers of CYP enzymes for 28 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/PD interaction with study drug.
  * Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
  * Hormone replacement therapy will also be allowed.
  * Subjects on a stable dose (at least 3 months) of thyroid medication will be allowed.
* An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (t) (AUC0-t) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.
Area under the concentration-time curve, from time 0 extrapolated to infinity (AUC0-inf) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.
Maximum observed concentration (Cmax) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.
Time to reach maximum observed concentration (Tmax) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.
Apparent terminal elimination rate constant (Kel) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.
Apparent terminal elimination half-life (T½) | 0 to 72 hours post dose
  The PK of MIV-711 following administration of single oral doses of capsule and tablet formulations under fasting and fed conditions in healthy subjects. The evaluation will be made between the formulations.

SECONDARY OUTCOMES:
The number and severity of AEs/SAE | from study start until 7+/-2 days after the last study drug administration
  Safety and tolerability of MIV-711 measured by number and severity of AEs/SAEs
The number of clinically significant abnormal lab results | from study start until 7+/-2 days after the last study drug administration
  Safety and tolerability of MIV-711 measured by number of clinical significant abnormal lab results.
The number of clinically significant ECG abnormalities | from study start until 7+/-2 days after the last study drug administration
  Safety and tolerability of MIV-711 measured by number of clinical significant ECG abnormalities.
The number of clinically significant physical examination abnormalities | from study start until 7+/-2 days after the last study drug administration
  Safety and tolerability of MIV-711 measured by number of clinical significant physical examination abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Hunt, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided